CLINICAL TRIAL: NCT04623580
Title: Flemish Inguinal and Femoral Hernia Prospective Registry
Acronym: FLIPR
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S59051
Record Dates: First submitted 2020-11-05; First posted 2020-11-10 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Herniorrhaphy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Inguinal or femoral hernia repair: All consecutive inguinal or femoral hernia repair (primary or mesh)
  Interventions: Device: Surgical inguinal or femoral hernia repair

INTERVENTIONS:
Device: Surgical inguinal or femoral hernia repair — Surgical inguinal or femoral hernia repair (primary or mesh)
  Other Names: Hernia repair

SUMMARY:
Prospective registry. The purpose of this clinical trial will be to measure surgical outcome parameters (e.g. recurrence, chronic pain and other quality indicators) after inguinal hernia repair using Patient Reported Outcome Measures (PROMs) in the short- and long-term.

DETAILED DESCRIPTION:
The primary objective is to investigate moderate to severe chronic pain 1 year after inguinal or femoral hernia repair, defined as numeric rating scale (NRS) ≥ 4, during daily activities.

The secondary objectives are:

* Surgical Site Occurrence (SSO) after 30 days
* Scope and incidence of pre- and postoperative pain (NRS 0 to 10)
* The difference between pre- and postoperative NRS scores (relative NRS score)
* Presence of pain and impact of pain on daily life activities
* Satisfaction and quality of life
* Sexual function
* Anxiety and depression
* Catastrophizing
* Recurrence
* Development of a predictive model for chronic pain.

ELIGIBILITY:
Inclusion criteria

* Consecutively all patients with a groin hernia (inguinal and/or femoral hernia) operated starting 01.01.2018.
* Male and female
* 18 years or older
* Operated of supervised by a participating surgeon (participating in this study is not necessarily by a whole surgical department of a hospital, but by specific surgeons)
* Elective and emergency surgery
* Primary and recurrent hernia
* Metachronous and synchronous hernia
* Signed informed consent form

Exclusion criteria

* Younger than 18 years
* Not operated or supervised by participating surgeon
* Pregnant at inclusion in the registry
* No signed informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: INGUINAL HERNIA PATIENTS
Sampling Method: Non-Probability Sample
Enrollment: 560 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Chronic pain after inguinal hernia repair | 5 years
  To investigate moderate to severe chronic pain 1 year after inguinal or femoral hernia repair, defined as numeric rating scale (NRS) ≥ 4, during daily activities.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - UZ Leuven, Leuven
  - Colette Barlé, Leuven